CLINICAL TRIAL: NCT05976776
Title: Effectiveness of a Childbirth and Parenthood Preparation Education on Maternal Health Needs, Pregnancy-Related Anxiety and Fetal Health Anxiety in Primigravidas
Brief Title: Effectiveness of a Childbirth and Parenthood Preparation Education in Primigravidas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Emine Akca, Assist. Prof. Dr. in the Amasya University Midwifery Department, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya Un
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related; Anxiety
Keywords: Maternal Health Needs; Fetal Health Anxiety; Primiparous women; Childbirth and Parenthood Preparation Education; Pregnancy-Related Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A randomized-controlled trial with pretest-posttest control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The Childbirth and Parenthood Preparation Education program
  Interventions: Behavioral: The Childbirth and Parenthood Preparation Education
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: The Childbirth and Parenthood Preparation Education — The "Childbirth and Parenthood Preparation Education" program will be applied to the experimental group for a period of 1 month (each week, once a week in total four sessions).
  Arms: Experimental group

SUMMARY:
To investigate the effect of the Childbirth and Parenthood Preparation Education on Maternal Health Needs, Pregnancy-Related Anxiety and Fetal Health Anxiety in Primigravidas. A total of 148 pregnant women are planned to be included in the study. Data will be collected with the 'Pregnant Identification Form', 'Maternal Health Needs Scale', 'Pregnancy-Related Anxiety Scale-Revision 2' and 'Fetal Health Anxiety Inventory. The "Childbirth and Parenthood Preparation Education" program will be applied to the experimental group for a period of four weeks (a month (each week, once a week in total four sessions)). It is thought that the results of the research will contribute to the welfare of pregnant women by reducing maternal health needs, pregnancy-related anxiety and fetal health anxiety levels.

DETAILED DESCRIPTION:
To investigate the effect of the Childbirth and Parenthood Preparation Education on Maternal Health Needs, Pregnancy-Related Anxiety and Fetal Health Anxiety in Primigravidas. A total of 148 pregnant women are planned to be included in the study. Data will be collected with the 'Pregnant Identification Form', 'Maternal Health Needs Scale', 'Pregnancy-Related Anxiety Scale-Revision 2' and 'Fetal Health Anxiety Inventory. The "Childbirth and Parenthood Preparation Education" program will be applied to the experimental group for a period of four weeks (a month (each week, once a week in total four sessions)). Within the scope of the "Childbirth and Parenthood Preparation training" program; Physiological and psychological changes in the mother during pregnancy, daily life during pregnancy, smoking, alcohol and substance use during pregnancy, exercise during pregnancy, nutrition and nutritional support during pregnancy, pregnancy follow-ups, routine examinations and immunization, common problems during pregnancy and suggestions for solutions, signs of danger during pregnancy and what to do, risky pregnancies, drug and human medicinal product management during pregnancy, labor process, drug-free methods for coping with labor pain, postpartum period and its characteristics, physiological changes in the mother after birth, psychological changes in puerperium, puerperal role and adaptation, postpartum behaviors , care of the newborn in the postpartum period, postpartum contraception methods will be explained. It is thought that the results of the research will contribute to the welfare of pregnant women by reducing maternal health needs, pregnancy-related anxiety and fetal health anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* 18-40 years old
* Primigravida
* Those who volunteered to participate in the research
* Pregnant women who do not have communication and mental difficulties

Exclusion Criteria:

* Those who do not fill out the entire questionnaire
* Those with risky pregnancy
* Pregnant women with a previous history of psychiatric illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 136 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Levels of Maternal Health Needs | 1 months
  Maternal Health Needs is one of the primary outcomes. This will be measured using 'Maternal Health Needs Scale (MHNS) '. The minimum score that can be obtained from the scale is "23", the maximum score is "115", and as the scale score increases, maternal health needs also increase.

SECONDARY OUTCOMES:
Pregnancy-Related Anxiety Levels | 1 months
  Pregnancy related anxiety level is another outcomes. This will be mesured using "Pregnancy-Related Anxiety Scale- Revision 2". The minimum score that can be obtained from the scale is "11", the maximum score is "55", as the score obtained from the scale increases, the level of anxiety in pregnancy also increases.
Fetal Health Anxiety Levels | 1 months
  Fetal Health Anxiety level is another outcomes. This will be mesured using "Fetal Health Anxiety Inventory (FHAI)". The minimum score that can be obtained from the scale is "0", the maximum score is "42", as the total score from the scale increases, the level of fetal health anxiety increases.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İbici Akça, Principal Investigator — Amasya University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minozzi S, Ambrosi L, Saulle R, Uhm SS, Terplan M, Sinclair JM, Agabio R. Psychosocial and medication interventions to stop or reduce alcohol consumption during pregnancy. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD015042. doi: 10.1002/14651858.CD015042.pub2. PMID 38682758